CLINICAL TRIAL: NCT02451371
Title: A Pilot Study for the Treatment of Refractory Auditory Verbal Hallucinations With Transcranial Direct Current Stimulation(tDCS) in Patients With Schizophrenia
Brief Title: Treatment of Refractory Auditory Verbal Hallucinations With tDCS in Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1501-022-638
Record Dates: First submitted 2015-04-27; First posted 2015-05-22 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Refractory auditory hallucination; tDCS
MeSH Terms: conditions — Schizophrenia; Hallucinations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tDCS (Experimental): Patients with schizophrenia to receive tDCS treatment
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — 2mA direct current, 20 minutes per session, 2 sessions per day with at least 3hours interval between sessions, a total of 10 tDCS sessions
  Other Names: YDT-201N

SUMMARY:
The purpose of this study is to exploratively evaluate the efficacy and safety of transcranial direct current stimulation (tDCS) in patients with schizophrenia who experience persistent auditory verbal hallucinations after adequate antipsychotics therapy for over three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia by the Diagnostic and Statistical Manual of Mental Disorders, Fourth edition, Text Revision (DSM-IV-TR)
* Presence of auditory hallucination after three months' trial of antipsychotics of adequate dose
* The Hamilton Program for Schizophrenia Voices Questionnaire (HPSVQ) score is at least 8

Exclusion Criteria:

* Significant brain pathology including head trauma, seizure, meningitis
* Intellectual disability (IQ < 70)
* Severe personality disorder
* Substance use disorder (except nicotine)
* Severe medical illness
* Disability in the sensory organs
* Pregnancy

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Auditory hallucination change by changes in The Psychotic Symptom Rating Scales (PSYRATs) Auditory hallucinations subscale score | approximately 2 weeks
  Auditory hallucination change by changes in the auditory hallucinations subscale from the Psychotic Symptom Rating Scales

SECONDARY OUTCOMES:
Electroencephalography - resting | approximately 2 weeks
  * change in lagged phase synchronization value
  * change in microstate connectivity value
Electroencephalography - P300 peak | approximately 2 weeks
  * change in P300 peak amplitude during auditory oddball task
  * change in P300 peak latency during auditory oddball task
Electroencephalography - P300 source | approximately 2 weeks
  * change in P300 source strength during auditory oddball task
  * change in P300 source location during auditory oddball task
Electroencephalography - P50 | approximately 2 weeks
  * change in T/C ratio (testing stimulus/conditioning stimulus) during paired click test
  * change in T/C difference (conditioning stimulus-testing stimulus) during paired click test
  * change in T/C difference (testing stimulus - conditioning stimulus) during paired click test
Electroencephalography - ERN (error-related negativity) peak | approximately 2 weeks
  * change in ERN peak amplitude during flanker task
  * change in ERN peak latency during flanker task
Electroencephalography - ERN (error-related negativity) source | approximately 2 weeks
  * change in ERN source strength during flanker task
  * change in ERN source location during flanker task
Electroencephalography - ERN (error-related negativity) frequency activity | approximately 2 weeks
  * change in ERN beta band activity during flanker task
  * change in ERN theta band activity during flanker task
  * change in ERN delta band activity during flanker task
Brain Magnetic Resonance Image (MRI) - T1 Image grey matter thickness | approximately 2 weeks
  change in grey matter thickness
Brain Magnetic Resonance Image (MRI) - T1 Image grey matter volume | approximately 2 weeks
  change in grey matter volume
Brain MRI - functional MRI | approximately 2 weeks
  change in Pearson's correlation coefficient of BOLD signals
Brain MRI - Diffusion Tensor Image (DTI) functional anisotropy | approximately 2 weeks
  change in fractional anisotropy
Brain MRI - Diffusion Tensor Image (DTI) mean diffusivity | approximately 2 weeks
  change in mean diffusivity
Brain MRI - Diffusion Tensor Image (DTI) radial diffusivity | approximately 2 weeks
  change in radial diffusivity
Brain MRI - Diffusion Tensor Image (DTI) axial diffusivity | approximately 2 weeks
  change in axial diffusivity
Brain MRI - myelin image | approximately 2 weeks
  change in myelin imaging intensity value
Kicer values change with treatment in striatum assessed by 18F-DOPA Positron Emission Tomography (PET) | approximately 2 weeks
  - Kicer values change with treatment in striatum
Magnetic Resonance Spectroscopy (MRS) | approximately 2 weeks
  - N-Acetyl Aspartate, Creatin, Choline, Myoinositol, Glutamate, Glutamine, GABA metabolite concentration change with treatment
Auditory hallucination change by changes in the Auditory Hallucination Rating Scale (AHRS) score | approximately 2 weeks
  Auditory hallucination change by changes in the Auditory Hallucination Rating Scale score
Auditory hallucination change by changes in the Korean Version of Hamilton Program for Schizophrenia Voices Questionnaire (HPSVQ) score | approximately 2 weeks
  Auditory hallucination change by changes in the Korean Version of Hamilton Program for Schizophrenia Voices Questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Jun Soo Kwon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea